CLINICAL TRIAL: NCT04105088
Title: Bayis Ilh Tus - A Strong Breath: Community-Based Research to Identify the Prevalence of and Contributors to Chronic Obstructive Pulmonary Disease in Remote and Rural First Nations Communities in British Columbia
Brief Title: Bayis Ilh Tus - A Strong Breath: Prevalence and Contributors to COPD in First Nations Communities in British Columbia
Acronym: ASB
Status: Recruiting | Type: Observational
Sponsor: University of British Columbia (Other)
Collaborators: Carrier Sekani Family Services (Unknown)
Responsible Party: Principal Investigator, Pat Camp, Associate Professor, University of British Columbia
Other Study IDs: ASB-2018
Record Dates: First submitted 2019-09-24; First posted 2019-09-26 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: First Nations; Indigenous; Epidemiology; Risk Factors; Community-based Research
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — dust samples from residences and community buildings
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Randomly-Sampled: Adults aged 30+ living in one of the First Nations communities whose household was randomly-sampled.
- Walk-in Volunteers: Adults aged 30+ living in one of the First Nations communities who is a walk-in study volunteer, not randomly-sampled.

SUMMARY:
Background. First Nations peoples in Canada carry an increased respiratory health burden compared to non-First Nations. However, there is little accurate information of how many First Nations people have COPD, especially in remote and rural areas.

Goal & Aims of the Study. The goal of this study is to estimate the burden of COPD in remote and rural First Nations communities. This project is a partnership between the University of British Columbia (UBC), Carrier Sekani Family Services (CSFS), and 13 First Nations communities in northern BC.

Aim 1: Estimate the prevalence of COPD and the magnitude of underdiagnosis. Aim 2: Characterize the relationship between inhaled pollutants (from residential, occupational, and community/cultural sources) and: 1) symptoms; 2) airflow obstruction; and 3) health care utilization.

Methodology. The investigators will recruit adults from randomly-selected households in 13 First Nations communities in northern BC. Detailed measurements of lung function, symptoms, self-reported exposure to lung irritants, air quality, and healthcare use will be collected.

Expected Outcomes. This study will provide an accurate estimate of the prevalence of COPD and, using a culturally-relevant community-based research approach, will identify the contribution of risk factors to COPD in First Nations communities.

DETAILED DESCRIPTION:
Background. First Nations peoples in Canada carry an increased respiratory health burden compared to non-First Nations. They are often exposed to high rates of indoor air pollution and cigarette smoke; and although there is a high use of acute health care services for chronic obstructive pulmonary disease (COPD), this disease is not "on the radar" in many First Nations communities. This may be because there is little accurate information of how many First Nations people have COPD, especially in remote and rural areas. The current estimates of prevalence of COPD in First Nations are based on self-report surveys, which are known to underestimate the true number threefold. Although it is well-known that cigarette smoking causes COPD, there has been less attention paid to the contribution of residential, historical/community/cultural, and occupational factors to the burden of COPD in First Nations people.

Goal & Aims of the Study. The goal of this study is to estimate the burden of COPD in remote and rural First Nations communities. This project is a partnership between the University of British Columbia (UBC), Carrier Sekani Family Services (CSFS), and 13 First Nations communities in northern BC.

Aim 1: Estimate the prevalence of COPD and the magnitude of underdiagnosis. Aim 2: Characterize the relationship between inhaled pollutants (from residential, occupational, and community/cultural sources) and: 1) symptoms; 2) airflow obstruction; and; 3) health care utilization.

The Primary Outcome is the prevalence of COPD.

Methodology. The investigators will recruit adults from randomly-selected households in 13 First Nations communities in northern BC. The investigators will collect detailed measurements of lung function, symptoms, self-reported exposure to lung irritants, and healthcare use. The investigators will also collect indoor air quality measures from homes and community buildings. For Aim 1, the prevalence and underdiagnosis of COPD will be estimated by measuring lung function using post-bronchodilator spirometry and comparing the presence of airflow obstruction with the diagnosis of COPD in the electronic health record. For Aim 2, the investigators will explore the relationship between inhaled indoor air pollutants and 1) current cough, wheeze, and dyspnea; 2) airflow obstruction; and 3) respiratory-related primary care visits or hospitalization, adjusting for age, sex, and smoking history.

Expected Outcomes. This study will provide an accurate estimate of the prevalence of COPD and, using a culturally-relevant community-based research approach, will identify the contribution of risk factors to COPD in First Nations communities. The Primary Outcome is the prevalence of COPD.

Significance of this Project. This project is a novel partnership between UBC, CSFS and partner Nations to explore the prevalence and risk factors of COPD, using a Indigenous approach to health research. This study is unique in being able to address the risks of COPD in remote and rural First Nations communities, which will lead to further work to identify strategies to reduce these risks and improve lung health.

ELIGIBILITY:
Inclusion Criteria:

* 30 years and older
* living in one of participating First Nations communities

Exclusion Criteria:

* confusion, dementia

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We will recruit members of the participating First Nations communities, aged 30 years and older.
Sampling Method: Probability Sample
Enrollment: 325 (Estimated)
Dates: Start 2018-02-13 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
forced expiratory volume, 1st second in litres | measured at study recruitment
  pre- and post-bronchodilator FEV1 to determine reversibility of airflow obstruction
forced vital capacity in litres | measured at study recruitment
  pre- and post-bronchodilator measures of vital capacity for use in the diagnosis of COPD
FEV1/FVC ratio | measured at study recruitment
  pre- and post-bronchodilator measures of FEV1/FVC to confirm diagnosis of COPD (where the FEV1 to FVC <0.70)

CONTACTS AND LOCATIONS:
Overall Officials: Pat G Camp, PhD, Principal Investigator — University of British Columbia; Travis Holyk, PhD, Study Director — Carrier Sekani Family Services
Locations (1):
- 13 individual First Nations in north-Central BC near Prince George, BC, Prince George, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No
No IPD is approved.

REFERENCES:
- [Derived] Turner J, Holyk T, Bartlett K, Rathburn B, Karlen B, Ervin F, Wilson J, Camp PG. "Bayis Ilh Tus - a strong breath" a community-based research project to estimate the prevalence of chronic obstructive pulmonary disease in remote and rural first nations communities in Canada: research protocol. Int J Equity Health. 2020 Jul 24;19(1):123. doi: 10.1186/s12939-020-01240-1. PMID 32709235